CLINICAL TRIAL: NCT04934436
Title: The Effect of Nursing Care Provided to Coronary Intensive Care Patients According to Their Circadian Rhythms on Sleep Quality, Pain, Anxiety and Delirium
Brief Title: The Effect of Nursing Care on Circadian Rhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Havva SERT, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAU
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Circadian Rhythm; Chronobiology Disorders; Biological Clock Disturbance; Nursing Care; Sleep Quality
MeSH Terms: conditions — Chronobiology Disorders; Sleep Initiation and Maintenance Disorders | interventions — Ear Protective Devices; Nursing Care

STUDY DESIGN:
Intervention Model Description: In terms of the reliability of the study results, the patients in this study will be allocated to the groups with a stratified randomization method. Patients will be randomly matched to the intervention (I) and control (C) group according to their gender, age, and circadian rhythms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): According to their chronotype, the intervention group will then be given sleeping glasses and earplugs at night for those who are in the morning type, and till afternoon during the day for those who are in the evening type. Moreover, patients in the intervention group will be given 5000 Lux daylight during the time they are awake depending on their circadian rhythms. An Android smartwatch will be used to determine patients' sleeping and waking up times, sleep quality and sleep depth. Nursing care will also be provided when patients are awake per their chronotype. Before the study, intensive care nurses will be trained to provide appropriate care according to the circadian rhythm and chronotype to have consistency in the care. Patients will be observed for three days and during this time cortisone and melatonin levels will be checked in both control and intervention groups. At the end of the third day, surveys will be conducted once again with both groups.
  Interventions: Other: sleeping glasses and earplug
- Control Group (No Intervention): All surveys that will be used in the study will be applied to both groups during the first and last interviews. The control group will not have any interventions, only the standard ICU care to be provided.

INTERVENTIONS:
Other: sleeping glasses and earplug — In this study, the effect of the chronotype-appropriate nursing care on the intervention group will be examined.
  Other Names: nursing care
  Arms: Intervention Group

SUMMARY:
The aim of this project is to determine the effect of nursing care provided to intensive unit care patients according to their circadian rhythms on sleep quality, pain, anxiety and delirium.

DETAILED DESCRIPTION:
During the current national and international literature review, the studies were seen to mostly focus on subjects such as circadian rhythm and psychological disorders and problems, obesity, cancer, etc. No studies were found on the effect of nursing care provided according to circadian rhythm. Therefore, it is thought that determining chronotypes and providing appropriate nursing care is important to prevent pain, sleep, delirium and many physiological parameters and comorbid diseases, especially in intensive care patients, in terms of maintaining the circadian rhythm.

The study population will consist of patients treated in the Coronary Intensive Care Unit of Sakarya University Training and Research Hospital. A total of 32 patients will form the sample of the study, including 16 in intervention and 16 in a control group that agree to participate in the study and meet the study criteria. In terms of the reliability of the study results, the patients in this study will be allocated to the groups with a stratified randomization method. Patients will be randomly matched to the intervention (I) and control (C) group according to their gender, age, and circadian rhythms. Data will be collected after obtaining the institution's permission, the approval of the Ethics Committee, and the patients' consent through a face-to-face interview with patients. Firstly, the patients will be evaluated after admitted to the intensive care unit, and the intervention and control group will be formed using a stratified randomized method from those meeting the study criteria. All surveys that will be used in the study will be applied to both groups during the first interview. According to their chronotype, the intervention group will then be given sleeping glasses and earplugs at night for those who are in the morningtype, and till afternoon during the day for those who are in the eveningtype. Moreover, patients in the intervention group will be given 5000 Lux daylight(Maldonado, 2017) during the time they are awake depending on their circadian rhythms. An Android smartwatch will be used to determine patients' sleeping and waking up times, sleep quality and sleep depth. Nursing care will also be provided when patients are awake per their chronotype. Before the study, intensive care nurses will be trained to provide appropriate care according to the circadian rhythm and chronotype to have consistency in the care. Patients will be observed for three days and during this time cortisone and melatonin levels will be checked in both control and intervention groups (this test is not provided regularly but it will be paid by the financial sponsors). At the end of the third day, surveys will be conducted once again with both groups. All through this time, the control group will not have any interventions, only the standard ICU care to be provided.

In the study, "Patient Information Form, The Richards-Campbell Sleep Questionnaire, the Sleep Quality Scale which is planned to be developed, Intensive Care Delirium Screening Checklist, Horne and Ostberg Morningness-Eveningness Questionnaire, Daily Rhythm Questionnaire, Hospital Anxiety and Depression Scale" will be used as a part of the pre-test. Three days later, "Patient Information Form, The Richards-Campbell Sleep Questionnaire, the Sleep Quality Scale which is planned to be developed, Intensive Care Delirium Screening Checklist, Horne and Ostberg Morningness-Eveningness Questionnaire, Daily Rhythm Questionnaire, Hospital Anxiety and Depression Scale" will be applied to the patients as a part of the post-test.

As part of this study, a new scale specific to intensive care patients will be developed. The effects of nursing care given in accordance with the circadian rhythm, which has not been investigated before, on sleep quality, pain, delirium, and anxiety will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being literate
* Not having communication difficulties (Sensory losses such as vision and hearing)
* Volunteering to participate in the research.
* Not having a psychiatric diagnosis by a specialist physician
* Being open to communication and cooperation
* Being admitted to the coronary intensive care unit due to Acute Coronary Syndrome and Myocardial Infarction

Exclusion Criteria:

* Having a diagnosed delirium
* Receiving ventilator support
* Using sleeping pills
* Having a diagnosis of dementia
* Insomnia/propensity to sleep as a side effect of the medication used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients will be randomly matched to the intervention (I) and control (C) group according to their gender, age, and circadian rhythms
Enrollment: 44 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the sleep quality | At the end of the 3rd day
  The effect of nursing care given in accordance with the chronotypes of individuals on sleep quality is the primary result for this study. This output measured by SQ-CC scale developed by authors.
Change in the pain levels | At the end of the 3rd day
  It was measured using VAS whether there was a decrease in the patients' pain scores as a result of the intervention after 3 days.
Change in the Anxiety levels | At the end of the 3rd day
  HADS was used to measure whether there was a decrease in the patients' anxiety levels as a result of the intervention after 3 days.
Change in the delirium score | At the end of the 3rd day
  After 3 days, it was measured using ICDSC whether the patients' rates of going into delirium decreased or whether their scores decreased as a result of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Meryem PELİN, Principal Investigator — Sakarya University Health Science Institute
Locations (1):
- Meryem PELİN, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelin M, Sert H. The effect of nursing care provided to coronary intensive care patients according to their circadian rhythms on sleep quality, pain, anxiety, and delirium: a randomised controlled trial. BMC Nurs. 2025 Feb 7;24(1):143. doi: 10.1186/s12912-025-02793-8. PMID 39920733